CLINICAL TRIAL: NCT03491969
Title: Clinical Study of Lipoic Acid on Ischemic Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xu Lei, Doctor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: LAoIHF
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Ischemic Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpha-Lipoic Acid(α-LA) (Experimental): Double blind treatment period consisted of treatment with CHF standard treatments, followed by α-LA 200 mg tid over a total duration of 24 months.
  Interventions: Drug: Alpha-Lipoic Acid(α-LA)
- Placebo (Placebo Comparator): Double blind treatment period consisted of treatment with CHF standard treatments, followed by Placebo 200 mg tid over a total duration of 24 months.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Alpha-Lipoic Acid(α-LA) — 200 mg, po, tid
  Arms: Alpha-Lipoic Acid(α-LA)
Drug: Placebos — 200 mg, po, tid
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy of alpha-lipoic acid(α-LA) on mortality in patients with ischemic heart failure (NYHA Class II - IV and EF =< 50%).

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years of age, male or female.

  * Patients with a diagnosis of AMI (>30 days) according to the global definition. ③Patients with a diagnosis of CHF (NYHA class II-IV) and reduced ejection fraction (EF =< 50%) and elevated BNP（NT-proBNP≥600pg/ml or BNP≥150pg/ml; NT-proBNP ≥400 pg/mL or BNP ≥100 pg/mL if patients was hospitalized for heart failure within 12months).

    * Patients must be treated with standardized heart failure medications treatment at a stable dose for at least 4 weeks.

      * Patients must give written informed consent before any assessment is performed.

Exclusion Criteria:

* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.

  * allergy to any of the study drugs, drugs of similar chemical classes（Vitamin B） as well as known or suspected contraindications to the study drugs.

    * Previous history of intolerance to recommended target doses of α-LA.

      * Current acute decompensated HF (exacerbation of chronic HF manifested by signs and symptoms that may require intravenous therapy).

        ⑤ Symptomatic hypotension and/or a SBP < 100 mmHg.

        ⑥ Severe liver function abnormalities (ALT or AST more than 3 times of the normal upper limit).

        ⑦ Estimated GFR < 30 mL/min/1.73m2 as measured by the simplified MDRD formula.

        ⑧ Serum potassium > 5.2 mmol/L.

        ⑨ Pregnant women or women preparing for birth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alpha-Lipoic Acid(α-LA) | Placebo
Started | 150 | 150
Completed | 138 | 139
Not Completed | 12 | 11

BASELINE CHARACTERISTICS:
Population: The primary efficacy endpoints were analyzed using the full analysis set (FAS), which followed the Intent-to-Treat (ITT) principle. Inclusion in the FAS required that participants receive the investigational drug for a minimum of 1 month. 300 patients were randomized in a 1:1 ratio to receive either ALA or a matching placebo. In the ALA group, 12 patients were excluded from the primary analysis. In the placebo group, 11 participants were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alpha-Lipoic Acid(α-LA) | Placebo | Total
Number analyzed (Participants) | 138 | 139 | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (10.7) | 65.7 (11.6) | 65.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 59
  Male | 108 | 110 | 218
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 138 | 139 | 277
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 138 | 139 | 277

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Had First Occurrence of the Composite Endpoint
Description: either all-cause death or heart failure (HF) hospitalization
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-Lipoic Acid(α-LA) | Placebo
Number analyzed (Participants) | 138 | 139
Participants | 32 | 40

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Alpha-Lipoic Acid(α-LA) | Placebo
All-Cause Mortality (participants affected / at risk) | 32/138 | 40/139
Serious Adverse Events (participants affected / at risk) | 12/145 | 14/144
Other Adverse Events (participants affected / at risk) | 31/145 | 25/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alpha-Lipoic Acid(α-LA) (N=145) | Placebo (N=144)
Death (General disorders) | 3 | 5
Hospitalization for Worsened heart failure (Cardiac disorders) | 4 | 7
Hospitalization for stroke (Nervous system disorders) | 3 | 1
Hospitalization for fracture (Injury, poisoning and procedural complications) | 1 | 1
Hospitalization for arterial occlusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alpha-Lipoic Acid(α-LA) (N=145) | Placebo (N=144)
Gastrointestinal symptoms (Gastrointestinal disorders) | 10 | 7
Infections (Infections and infestations) | 11 | 12
Worsened renal function (Renal and urinary disorders) | 7 | 4
Dizziness (Nervous system disorders) | 3 | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT03491969/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03491969/SAP_001.pdf